CLINICAL TRIAL: NCT04206631
Title: Effectiveness of Comedone Extraction and Oral Doxycycline In The First Line Treatment of Moderate Acne Vulgaris: Study on HIF-1 Alpha Expression
Brief Title: Comedone Extraction and Oral Doxycycline In The First Line Treatment of Moderate Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr.dr.Irma Bernadette, SpKK (K), Irma Bernadette S. Sitohang, MD, PhD - Head of Division of Cosmetic Dermatology, Department of Dermatology and Venereology, Faculty of Medicine, Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ComExt
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Acne Vulgaris
Keywords: comedone extraction; oral doxycycline; moderate acne vulgaris; HIF-1 alpha expression
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycycline Group (Placebo Comparator): Subjects were randomized to receive Doxycycline capsules. The capsules were taken once daily for 6 weeks and evaluated every 2 weeks.
  Interventions: Drug: Doxycycline Capsule
- Comedone Extraction Group (Active Comparator): Subjects were randomized to receive comedone extraction. Comedone extraction were done three times, and evaluated every 2 weeks.
  Interventions: Procedure: Comedone extraction

INTERVENTIONS:
Drug: Doxycycline Capsule — Doxycycline capsule 100 mg/day, tretinoin cream 0.05% on face every night, benzoyl peroxide gel 2.5% on face in the morning and afternoon.
  Arms: Doxycycline Group
Procedure: Comedone extraction — Comedone extraction, tretinoin cream 0.05% on face every night, benzoyl peroxide gel 2.5% on face in the morning and afternoon.
  Arms: Comedone Extraction Group

SUMMARY:
The objective of the study was to evaluate the effectiveness of comedone extraction compared to oral antibiotics as the main therapy of moderate acne vulgaris (MAV); and to determine the expression of HIF-1 alpha by examining the immunohistochemistry and ELISA as a sign of hypoxia/anoxia in MAV lesion. This was a randomized, placebo-controlled clinical trial that was performed in 2015 at three different dermatology clinics in Indonesia, Cipto Mangunkusumo Hospital Jakarta, Gatot Soebroto Army Hospital Jakarta, and PT. Mattel Indonesia, Cikarang. One hundred and twenty eight subjects with moderate acne vulgaris were recruited and randomized to receive either oral doxycycline or comedone extraction for six weeks. Subjects who had acne lesion and the back area were offered skin lesion biopsy to evaluate immunohistochemistry and ELISA before administration of medication. The main outcome was total reduction of inflammatory and non inflammatory lesions, evaluated every two weeks.

DETAILED DESCRIPTION:
Acne vulgaris (AV) is a polymorphic disease, characterized by inflammatory and noninflammatory lesions. Systemic antibiotics play a role as the first line therapy of moderate acne vulgaris treatment. Since bacterial resistance tends to increase, alternative therapy for moderate acne vulgaris is needed.

This study aims to evaluate the effectiveness of comedone extraction compared to oral antibiotics as the main therapy of moderate acne vulgaris; and to etermine the expression of HIF-1 alpha by examining the immunohistochemistry and ELISA as a sign of hypoxia/anoxia in MAV lesion.

This was a randomized, placebo-controlled clinical trial that was performed in 2015 at three different dermatology clinics in Indonesia, Cipto Mangunkusumo Hospital Jakarta, Gatot Soebroto Army Hospital Jakarta, and PT. Mattel Indonesia, Cikarang.

One hundred and twenty eight subjects, aged between 15 and 50 years, with moderate acne vulgaris were recruited and randomized to receive either oral doxycycline (100 mg) or comedone extraction for six weeks. Subjects who had acne lesion and the back area were offered skin lesion biopsy to evaluate immunohistochemistry and ELISA before administration of medication.

At each follow-up visit, subjects were asked to grade the overall response and questioned regarding adverse events. The objective or main outcome was total reduction of inflammatory and noninflammatory lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate acne vulgaris based on clinical manifestation of face (20-100 comedones, 15-50 inflammatory lesions, and/or 30-125 total lesions)
* Age range of 15 to 50 years old

Exclusion Criteria:

* History of oral antibiotics consumption within 2 weeks preceding this study
* Usage of topical retinoid in less than previous 2 weeks
* History of systemic retinoid consumption within 3 months preceding this study
* Pregnant of breastfeeding women
* Consuming oral contraception during examination
* Drug allergy or skin manifestation due to side effect of moderate acne vulgaris first line therapy

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-10-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Inflammatory Lesions at 2 weeks | 2 weeks
  Numeric data of total reduction (improvement) of inflammatory lesions
  (Baseline inflammatory lesion count) - (Week 2 inflammatory lesion count)
  __________________________________________________________ x 100% Baseline inflammatory lesion count
Change from Baseline Inflammatory Lesions at 4 weeks | 4 weeks
  Numeric data of total reduction (improvement) of inflammatory lesions
  (Baseline inflammatory lesion count) - (Week 4 inflammatory lesion count)
  __________________________________________________________ x 100% Baseline inflammatory lesion count
Change from Baseline Inflammatory Lesions at 6 weeks | 6 weeks
  Numeric data of total reduction (improvement) of inflammatory lesions
  (Baseline inflammatory lesion count) - (Week 6 inflammatory lesion count)
  __________________________________________________________ x 100% Baseline inflammatory lesion count
Change from Baseline Non-Inflammatory Lesions at 2 weeks | 2 weeks
  Numeric data of total reduction (improvement) of non-inflammatory lesions
  (Baseline non-inflammatory lesion count) - (Week 2 non-inflammatory lesion count)
  __________________________________________________________ x 100% Baseline non-inflammatory lesion count
Change from Baseline Non-Inflammatory Lesions at 4 weeks | 4 weeks
  Numeric data of total reduction (improvement) of non-inflammatory lesions
  (Baseline non-inflammatory lesion count) - (Week 4 non-inflammatory lesion count)
  __________________________________________________________ x 100% Baseline non-inflammatory lesion count
Change from Baseline Non-Inflammatory Lesions at 6 weeks | 6 weeks
  Numeric data of total reduction (improvement) of non-inflammatory lesions
  (Baseline non-inflammatory lesion count) - (Week 6 non-inflammatory lesion count)
  __________________________________________________________ x 100% Baseline non-inflammatory lesion count

SECONDARY OUTCOMES:
Subjective Improvement at 2 weeks | 2 weeks
  Improvement of clinical manifestation based on subjective complaints. Subjects were asked to grade overall response using rating scale (0-4), with higher score means a better outcome (0) no or minimal improvement
  1. mild improvement
  2. moderate improvement
  3. robust improvement
  4. very good improvement
Subjective Improvement at 4 weeks | 4 weeks
  Improvement of clinical manifestation based on subjective complaints. Subjects were asked to grade overall response using rating scale (0-4), with higher score means a better outcome (0) no or minimal improvement
  1. mild improvement
  2. moderate improvement
  3. robust improvement
  4. very good improvement
Subjective Improvement at 6 weeks | 6 weeks
  Improvement of clinical manifestation based on subjective complaints. Subjects were asked to grade overall response using rating scale (0-4), with higher score means a better outcome (0) no or minimal improvement
  1. mild improvement
  2. moderate improvement
  3. robust improvement
  4. very good improvement
Number of Participants with Side Effects at 2 weeks | 2 weeks
  * Mild side effects if it did not need further management and research medication could be continued.
  * Moderate side effects if clinical manifestations were robust, itchy, pain, erythematous, yet did not need further management and temporary.
  * Severe side effects if it interfered daily activity, such as burn and pain sensastion, erythematous skin, edema, skin exfoliation, that needed further management.
Number of Participants with Side Effects at 4 weeks | 4 weeks
  * Mild side effects if it did not need further management and research medication could be continued.
  * Moderate side effects if clinical manifestations were robust, itchy, pain, erythematous, yet did not need further management and temporary.
  * Severe side effects if it interfered daily activity, such as burn and pain sensastion, erythematous skin, edema, skin exfoliation, that needed further management.
Number of Participants with Side Effects at 6 weeks | 6 weeks
  * Mild side effects if it did not need further management and research medication could be continued.
  * Moderate side effects if clinical manifestations were robust, itchy, pain, erythematous, yet did not need further management and temporary.
  * Severe side effects if it interfered daily activity, such as burn and pain sensastion, erythematous skin, edema, skin exfoliation, that needed further management.

OTHER OUTCOMES:
Expression of Antibody HIF-1 Alpha with Immunohistochemistry Examination | Baseline
  Analysis of HIF-1 Alpha expression on keratinocyte cell of pilosebaceous ducts (samples from skin lesion biopsy) was examined with immunohistochemistry using antibody HIF-1 alpha which was visualized with microscope and photographed to achieve qualitative data.
Expression of Antibody HIF-1 Alpha with ELISA Examination | Baseline
  The measurement of HIF-1 Alpha protein concentration in the sebaceous follicle ducts was conducted through ELISA examination with Cusabio Human Hypoxia-inducible factor

CONTACTS AND LOCATIONS:
Overall Officials: Irma B Sitohang, MD, PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sitohang IBS, Soebaryo RW, Kanoko M. Acne Lesion Extraction versus Oral Doxycycline for Moderate Acne Vulgaris: A Randomized Clinical Trial. J Clin Aesthet Dermatol. 2021 Jun;14(6):E61-E65. Epub 2021 Jun 1. PMID 34804358